CLINICAL TRIAL: NCT05966220
Title: Post Market Clinical Follow-up of Hip Surgery Using FH ORTHO Company Medical Devices (FH ORTHO Company Hip Observatory).
Brief Title: Post Market Clinical Follow-up of Hip Surgery Using FH ORTHO Company Medical Devices.
Acronym: HipFHOrtho
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FH ORTHO (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-01
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hip Surgery
Keywords: hip prosthesis, observatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total hip arthroplasty (THA) and Revision THA (Other): Patients will be monitored for up to 15 years postoperatively.
  Interventions: Device: Hip surgery with FH Ortho devices
- Traumatology: femoral neck Total hip arthroplasty or hemiarthroplasty (Other): Patients will be monitored for up to 10 years postoperatively.
  Interventions: Device: Hip surgery with FH Ortho devices

INTERVENTIONS:
Device: Hip surgery with FH Ortho devices — This study is a real-life observatory designed to collect long-term clinical data on patients who have undergone hip joint replacement or repair following hip trauma.
  In this type of intervention, one or more medical devices distributed by FH ORTHO Company may be used by surgeons.

SUMMARY:
The objective of this observatory is to generate additional real life clinical data in accordance with local regulation (i.e. Post-Market Clinical Follow-up (PMCF) study, a study carried out following the European Conformity (CE) marking of a device and intended to answer specific questions relating to clinical safety or performance (i.e. residual risks) of a device when used in accordance with its approved labelling).

The difficulty of such an observatory is to be able to collect data on the different versions of the devices, on the different possible combinations of implants of an arthroplasty. The observatory must also be able to cover devices used in surgery to repair osteoarticular trauma.

The observatory will be based on the principle of a "dynamic" cohort during the inclusion period, i.e. with possible inclusions to replace the premature exits.

Technical solutions will be implemented to facilitate data collection from surgeons (electronic Case Report Form (eCRF) and from patients (Electronic Patient Reported Outcome (ePRO) on phone/tablet/computer).

ELIGIBILITY:
Inclusion Criteria:

1. Any patient undergoing or having undergone implantation of medical devices distributed by FH ORTHO Company for hip arthroplasty and traumatology, used in accordance with their approved Instruction For Use, in one of the centers participating in the Observatory.
2. Patient is at least 18 years of age.
3. Patient agreeing to participate after having been informed orally and in writing (with written consent if required locally).
4. In some countries, such as France, the patient will have to be socially insured to be included in the study.

Exclusion Criteria:

1. An infection, or latent infection.
2. A mental or neuromuscular disorder that would create an unacceptable risk of prosthetic instability, failure of prosthetic fixation, or post-operative complications (except for the HIP&GO Double mobility cemented cup and, if applicable, the associated stems and heads when assembled together).
3. Known Insufficient bone quality and/or bone stock.
4. Known allergy to any component of the material listed on the product label.
5. Metabolic diseases that could compromise bone regrowth.
6. Metabolic and/or vascular treatment or disease that may compromise bone healing or consolidation.
7. Drug dependency.
8. Uncooperative patient unable to follow recommendations.
9. Protected adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2038-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate (revision) of the medical device over the long term (maximum 15 years). | maximum 15 years.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Clinique Pasteur, Guilherand-Granges
  - Centre Hospitalier Du Haut Bugey, Oyonnax
  - Polyclinique Reims-Courlancy, Reims
  - Clinique Mutualiste La Sagesse, Rennes
  - Clinique de l'Atlantique, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No